CLINICAL TRIAL: NCT04669028
Title: A Phase 3, Double Blind, Randomized, Placebo Controlled, Parallel Group, Multicenter Study of NE3107 in Subjects Who Have Mild to Moderate Probable Alzheimer's Disease
Brief Title: A Phase 3 Study of NE3107 in Probable Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM101
Record Dates: First submitted 2020-12-04; First posted 2020-12-16 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NE3107 (Experimental): Hard gelatin capsule containing 20 mg micronized NE3107 drug substance blended with common excipients for oral formulations
  Interventions: Drug: NE3107
- placebo (Placebo Comparator): Hard gelatin capsule containing only common excipients for oral formulations
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NE3107 — NE3107 is an investigational orally bioavailable, blood-brain barrier permeable anti-inflammatory agent with a new mechanism of action targeting multiple mechanisms of pathology in Alzheimer's disease.
  Arms: NE3107
Drug: Placebo — capsules that do not contain NE3107
  Arms: placebo

SUMMARY:
U.S. multicenter, parallel group study designed to evaluate the safety and efficacy of oral 20 mg twice daily (BID) NE3107 vs placebo in 400 adult subjects with mild to moderate probable AD. Dual co-primary endpoints (Clinical Dementia Rating Scale Sum of Boxes, CDR-SB and ADAS-Cog12) will be evaluated as the change from Baseline to Week 30. Secondary endpoints include measures of cognition, neuropsychological deficits, functional performance, and glycemic control. A subset of patients may volunteer for exploratory magnetic resonance imaging (volumetric changes) and positron emission tomography (cortical glucose metabolic rate) scans at baseline and week 30.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female subject aged 60 to 85 y at Screening (V1). 2. Has mild to moderate probable AD as defined by all of the following criteria:

  1. Meets the National Institute on Aging and Alzheimer's Association (NIA-AA, 2011) criteria of all cause dementia and probable AD.
  2. Has a Clinical Dementia Rating (CDR) (Section 8.1.6) Standard Global Score of 1 to 2, inclusive (mild to moderate).
  3. Has a MMSE score of ≥14 and ≤24 at both Screening and Baseline visits. The difference in scores between Screening and Baseline must be < 3 points (i.e., the difference must not exceed 3 points). (Section 8.1.5)
  4. Has an historical MRI or CT scan of the brain on file no earlier than AD diagnosis that fails to exhibit features of another potential pathobiology that could better account for the cognitive disorder.

     3. Historical evidence of impairment on a mental status exam or documented prior diagnosis of or treatment for dementia from a health care professional.

     4. Has a modified Hachinski Ischemic Scale (Section 8.1.8) score of ≤4 at Screening (V1).

     5. If taking an anticholinesterase inhibitor (AChEI) (e.g., donepezil, galantamine, rivastigmine) and/or memantine at Screening (V1):

  <!-- -->

  1. Must have been taking the medication(s) for ≥3 mo, and
  2. Current dose regimen and form must have remained stable for ≥6 wk and must remain stable throughout participation in the study.

     NOTE: Subjects not being treated with an AChEI and/or memantine at Screening (V1) may also be enrolled if initiation of an AChEI and/or memantine is not planned for the time period during which the subject will be participating in this study.

     NOTE: Dosage changes during the study due to clinical deterioration should be discussed with the Medical Monitor prior to being implemented.

     6. If taking medications for glycemic control at the time of Screening (V1), must be stable on the current dose regimen and form for ≥3 mo prior to randomization and must remain stable throughout participation in the study.

     7. Females taking hormone replacement therapy (HRT) must have maintained a stable regimen for at least two years prior to randomization and agree to continue the regimen until completing the final safety assessment in Week 30 at the end of the study.

     8. Must meet one of the following criteria:

  <!-- -->

  1. Females: Surgically sterilized (e.g., hysterectomy, bilateral oophorectomy, or tubal ligation) for at least 6 mo prior to Screening (V1) or postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 y; if needed, the Investigator may confirm menopausal status through an FSH assessment at Screening [V1]). 6.8.1
  2. Males: Vasectomized. If not vasectomized, must use an appropriate contraception method as noted in Section 6.8.1.

     9. Must provide voluntary written informed consent prior to Screening (V1). If the subject is unable to provide informed consent due to cognitive status, the subject must provide assent and a legally authorized representative provides full written informed consent on behalf of the subject.

     10. Willing to allow collection of blood for ApoE genotyping. 11. Able to comply with the study procedures, in the opinion of the Investigator.

     12. Has a primary caregiver/study partner willing to accept responsibility for supervising the treatment (e.g., administering study drug), accompanying the subject to clinic visits and assessing the condition of the subject throughout the study in accordance with all protocol requirements. The primary caregiver/study partner must be willing to sign the caregiver ICF.

     Exclusion Criteria:
* 1. Has prior brain imaging inconsistent with probable AD 2. A history of a stroke that resulted in a cognitive or motor deficit or, MRI or CT evidence of a moderate or large cerebral infarct.

  1. Should there be any evidence of neurologic symptoms between the date of the scan confirming diagnosis and Screening (V1), rescanning is necessary.

     3. Has clinically relevant abnormal laboratory tests including serum vitamin B12 deficiency, thyroid function abnormality, severe anemia, or electrolyte abnormality.

     4. Diagnosis of type 1 diabetes or type 2 diabetes requiring insulin treatment or the need to use continuous glucose monitoring. Subjects who become insulin dependent during the study may not continue to participate in the study.

     5. History of epilepsy or seizure disorder requiring ongoing treatment, or any seizure or loss of consciousness within 12 mo prior to Screening (V1).

     6. Subjects are ineligible, if in the opinion of the investigator, they have deficits in speech, comprehension, auditory functioning, or vision which would adversely impact their ability to perform the study's cognitive test procedures, complete rating scales, or engage in interviews.

     7. Has any of the following laboratory findings at Screening (V1):

  <!-- -->

  1. Alanine aminotransferase >3 × upper limit of normal (ULN), aspartate aminotransferase >3 × ULN, or history of clinically significant liver disease in the Investigator's medical judgment.
  2. Hemoglobin ≤10 g/dL.
  3. International normalized ratio >1.5 if not on anticoagulant medication; if the subject is on anticoagulant medication, the anticoagulant medication should be optimized and on a stable dose for ≥4 wk prior to Screening (V1).
  4. Creatinine clearance (Cockcroft Gault formula) of <45 mL/min.
  5. Known to be seropositive for human immunodeficiency virus (1 and 2), hepatitis B, or hepatitis C. Subjects with hepatitis C who had spontaneous resolution or received successful curative treatment (e.g., HARVONI® [ledipasvir/sofosbuvir]) with a documentation of undetectable viral load for at least 3 mo may be allowed. Serological testing will not be performed as part of this study.

     8. Female subjects with child-bearing potential (premenopausal, menstrual bleeding within the last 12 months) or who are pregnant or breastfeeding.

     9. History of any medical illness such as cancer requiring systemic therapy in the last 5 y, except for localized basal cell carcinoma of the skin, in situ cervical cancer successfully treated with surgical excision, and stable (for ≥90 d prior to Screening [V1]) prostate cancer.

     10. History of breast cancer. 11. History of severe heart failure (Grade 2 or higher on the New York Heart Association scale), major stroke, uncontrolled seizure disorder, or other medical illness that, in the Investigator's opinion, will increase the subject's risk of participation in the study or confound study assessments.

     12. Any surgery requiring general anesthesia that is planned to occur during the study. Local anesthesia during outpatient surgery is permitted if, in the opinion of the Investigator, the operation will not interfere with study procedures and subject safety.

     13. History or current evidence of major psychiatric illness such as schizophrenia, bipolar disorder, or major depressive disorder that may interfere with the subject's ability to perform the study and all assessments.

  <!-- -->

  1. Geriatric Depression Scale Short Form (GDS SF) score >8 at Screening (V1). NOTE: Mild depression or depressive mood arising in the context of AD are not criteria for exclusion. The use of anti epileptic medication for non-seizure-related treatment or the use of antidepressants is allowed if the dose has remained stable for ≥60 d prior Screening (V1).

     14. Violent or aggressive behavior that may interfere with study participation 15. History of active suicidal thoughts (Type 4 or 5 on the C SSRS) in the 6 mo prior to Screening (V1) or at Baseline (V2), history of a suicide attempt in the previous 2 y or >1 lifetime suicide attempt, or are at serious suicide risk, in the Investigator's clinical judgment.

     16. History of alcohol or drug abuse or dependence within 24 mo of Screening (V1) as defined by the Diagnostic and Statistical Manual of Mental Disorders 5.

  <!-- -->

  1. Positive urine screen for drugs of abuse that include methadone, cocaine, and amphetamines; positive urine screen for opiates, barbiturates, or benzodiazepines without a prescription.

     17. Has participated in another Investigational New Drug research study involving small molecule drugs within 60 d or biological drugs within 90 d prior to the first dose of study drug in this study (Baseline [V2]) or within 5 half-lives of the other investigational medicinal product, whichever is longer.

     18. History of Covid-19 (SARS-CoV-2) infection within 6-weeks prior to screening. Subjects with unresolved symptoms of Covid-19 infection or ongoing cognitive or other deficits attributable to post-Covid-19, that may affect participant safety or interfere with efficacy assessments, based on the Investigator's clinical judgment.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) | baseline and week 30 (end of study)
  test of 6 cognitive or functional domains, including memory, orientation, judgment, community affairs, home hobbies, and personal care are scored by certified raters after interviewing both participants and their informants. Higher score is indicative of more severe disease. The minimum score is 0 and the maximum score is 18. The CDR-SB is a co-primary outcome with ADAS-Cog12
Change in Alzheimer's Disease Assessment Scale Cognitive Subscale 12 [ADAS Cog12] | baseline and week 30 (end of study)
  The ADAS-Cog was developed to assess the level of cognitive dysfunction in Alzheimer's disease. It is also used in studies of interventions in people with mild cognitive impairment. It is also used for assessing the efficacy of antidementia treatments. The test is administered and scored by a certified rater to assess the cognitive domains of memory, language, orientation and praxis. A higher score is indicative of more severe disease, with 0 (no cognitive deficit) being the lowest score possible and 80 being the highest score and associated with severe cognitive impairment. ADAS-Cog12 is a co-primary outcome with CDR-SB.

SECONDARY OUTCOMES:
Alzheimer's Disease clinical COMposite Score (ADCOMS) | baseline and week 30 (end of study)
  composite score of questions from different cognitive tests (CDR, MMSE, and ADAS-Cog12). total score ranges from 0-1.97, with higher scores indicating worse disease
Alzheimer's Disease Cooperative Study Activities of Daily Living Scale | baseline and week 30 (end of study)
  23 item scale with total score of 0-78, with a lower score indicating worse disease
Mini Mental State Exam (MMSE) | baseline and week 30 (end of study)
  30 questions with a total score of 0-30, with a lower score indicating worse disease
Alzheimer's Disease Cooperative Study Clinical Global Impression of Change [ADCS CGIC] | baseline and week 30 (end of study)
  The ADCS-CGIC focuses on clinicians' observations of change in the subject's cognitive, functional, and behavioral performance since the beginning of a trial. It relies on both direct examination of the subject and interview of informants (e.g. trial partner). global severity at baseline scored from 1 (normal, not at all ill) to 7 (among the most extremely ill patients); and global change at follow-up scored from 1 (marked improvement) to 7 (marked worsening), where 4 indicates no change.
Neuropsychiatric Index 12 | baseline and week 30 (end of study)
  12 questions with total score 0-12, with higher score indicating worse disease
CDR Global Score | baseline and week 30 (end of study)
  The CDR is a 5-point scale used to characterize 6 domains of cognitive and functional performance applicable to AD and related dementias. Higher score is more severe disease symptoms. The overall CDR Global Score is calculated through the use of an algorithm. 0= normal, 0.5= very mild dementia, 1=mild dementia, 2=moderate dementia, 3=severe dementia

OTHER OUTCOMES:
Resource Utilization in Dementia (short version, Lite) | baseline and week 30 (end of study)
  compiles data on the use of social services, frequency and duration of hospitalizations, unscheduled contacts with health care professionals, use of concomitant medications by both the caregiver and the patient, amount of time the caregiver spends caring for the patient and missing work, and patients' use of study medication.
volumetric magnetic resonance imaging (vMRI) | baseline and week 30 (end of study)
cortical metabolic rate using fluorodeoxyglucose positron emission | baseline and week 30 (end of study)
fasting blood glucose | baseline and week 30 (end of study)
  measures glucose concentration in blood after overnight fasting
postprandial glucose excursions | baseline and week 30 (end of study)
  3-day average of postprandial glucose measure by continuous glucose monitoring
Homeostatic assessment of insulin resistance 2 (HOMA2-IR) | baseline and week 30 (end of study)
  blood tests for insulin and glucose levels
C-reactive protein | baseline and week 30 (end of study)
  blood test
plasma ratio of amyloid beta 1-42/1-40 | baseline and week 30 (end of study)
  blood test
plasma concentration of phospho-tau 217 | baseline and week 30 (end of study)
  blood test
plasma concentration of glial fibrillary acidic protein | baseline and week 30 (end of study)
  blood test
plasma concentration of Neurofilament light (NfL) | baseline and week 30 (end of study)
  blood test
change in DNA methylation of genes associated with measures of biological age | baseline and week 30 (end of study)
  blood test
change concentration of serum leptin | baseline and week 30 (end of study)
  blood test
change in concentration of serum adiponectin | baseline and week 30 (end of study)
  blood test
change in plasma concentration of tumor necrosis factor (TNF) | baseline and week 30 (end of study)
  blood test
change in plasma concentration of monocyte chemoattractant protein (MCP1) | baseline and week 30 (end of study)
  blood test

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reading CL, Ahlem CN, Murphy MF. NM101 Phase III study of NE3107 in Alzheimer's disease: rationale, design and therapeutic modulation of neuroinflammation and insulin resistance. Neurodegener Dis Manag. 2021 Aug;11(4):289-298. doi: 10.2217/nmt-2021-0022. Epub 2021 Jul 12. PMID 34251287
- [Derived] Reading CL, Yan J, Testa MA, Simonson DC, Javaid H, Schmunk L, Martin-Herranz DE, Brooke R, Gordevicius J, Zhang J, Yuan H, Ahlem C, Wang L, Markham P, Osman N, O'Quinn S, Palumbo J. An exploratory analysis of bezisterim treatment associated with decreased biological age acceleration, and improved clinical measure and biomarker changes in mild-to-moderate probable Alzheimer's disease. Front Neurosci. 2025 May 2;19:1516746. doi: 10.3389/fnins.2025.1516746. eCollection 2025. PMID 40386807